CLINICAL TRIAL: NCT05437822
Title: Effect of Tranexamic Acid in Proximal Humeral Fracture Surgery. A Randomized Controlled Trial
Brief Title: Tranexamic Acid in Proximal Humeral Fractures
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Elda University Hospital (Other)
Collaborators: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, Alejandro Lizaur-Utrilla, PhD, MD, Head of Orthopaedic Surgery Department, Elda University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TXA-Humeral Fracture
Record Dates: First submitted 2022-06-18; First posted 2022-06-29 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Proximal Humeral Fracture; Surgical Treatment
Keywords: proximal humeral fracture; surgical treatment; Tranexamic acid
MeSH Terms: conditions — Shoulder Fractures | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: All patients will be treated surgically with an internal fixation or arthroplasty. The two patient groups will include: 1) Study group treated with topic tranexamic acid infused in shoulder joint; 2) Control group with no drug treatment.
  Blood transfusion criteria will remain consistent with hospital standards. Deep vein thrombosis (DVT) prophylaxis will remain consistent with hospital standards (subcutaneous heparin from admission until 12 hours prior to surgery and beginning 6 hours after surgery).
  Patients will be followed 30 days
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will be allocated into two groups based on randomized 20-block method by an independent assistant using computer generated randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TXA group (Experimental): Tranexamic acid, a topic dose of 2 g diluted in 50 mL saline solution infused in shoulder joint
  Interventions: Drug: Tranexamic acid
- Control group (No Intervention): In the control group will not be administered TXA or any other drugs.

INTERVENTIONS:
Drug: Tranexamic acid — 2 g of tranexamic acid in 50 mL of saline
  Arms: TXA group

SUMMARY:
The purpose of this study is to determine the effect of tranexamic acid (on blood loss and transfusion requirements in patients with proximal humeral fractures requiring open surgical approaches.

This a blinded, controlled, therapeutic trial in which the patients will be randomized to receive TXA or no drug intervention. The primary outcome is the estimated total blood loss.

This study presents only minimal risks for the included patients.

DETAILED DESCRIPTION:
Studies have shown that hip fractures have a significant perioperative blood loss. Postoperative anaemia is associated with a higher morbidity and mortality.

Tranexamic acid is a safe and effective antifibrinolytic widely used to reduce blood loss in other forms of orthopaedic surgery and in traumatized patients. However, evidence on the effectiveness of TXA in shoulder fractures is more limited. Proximal humeral fractures represent a common orthopedic injury in elderly patients The goal of this study is to assess if the use of topic tranexamic acid in patients with proximal humeral fractures will result in a reduction in blood losses and blood transfusion rates.

The hypothesis is that by providing topic TXA at the end of surgery will decrease the amount of preoperative and intraoperative bleeding thereby leading to a decreased need for postoperative transfusion.

This a blinded, controlled, therapeutic trial in which the patients will be randomized to receive TXA or no drug intervention. The primary outcome is the estimated total blood loss. Secondary outcomes, need for blood transfusion, length of stay, and rate of thromboembolic events.

Candidates for the study will be consecutive patients with a diagnosis of proximal humeral fracture. All patients meeting inclusion criteria will be recruited for enrollment into the study. Informed consent will be obtained from the patient prior to randomization.

At that time, each patient will be randomized into one of two groups by an independent staff using computer generated randomization and allocation concealment. The two patient groups will include:

1. Study group: 2 g of tranexamic acid topically infused in shoulder joint before surgical closure.
2. Control group: no intervention Both patient groups will be blinded with regard to drug intervention. Patients will be treated surgically with internal fixation or arthroplasty. Blood transfusion criteria will remain consistent with hospital standards (Hb<7 g/dL or >9 g/dL if symptomatic anemia). Total number of blood transfusions received will be documented upon patient discharge.

Deep vein thrombosis (DVT) prophylaxis will remain consistent with hospital standards (subcutaneous heparin from admission until 12 hours prior to surgery and beginning 6 hours after surgery).

Patients will be followed 30 days. Diagnostic studies to assess for thromboembolic events (i.e. DVT, pulmonary embolism (PE), and stroke) will be ordered only if the patient develops clinical signs or symptoms that justify their use.

ELIGIBILITY:
Inclusion Criteria:

* Acute proximal humeral fracture
* Age over 18 years

Exclusion Criteria:

* ASA IV
* Concomitant fracture
* Refusal to receive blood products
* Allergy for tranexamic acid
* Severe hepatic dysfunction (AST/ALT >60)
* Renal function impairment (serum creatinine > 2 mg/dL or creatinine clearance <30 mL/min),) or kidney transplant
* Active acute thromboembolic event in the past 12 months (Deep Vein Thrombosis, Pulmonary)
* Active coronary artery disease or cerebrovascular accident (event in the past 12 months).
* Coronary stents
* History of hypercoagulability
* Coagulopathy (INR > 1.4)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-29 (Actual); Primary Completion 2023-06-21 (Estimated); Study Completion 2023-06-24 (Estimated)

PRIMARY OUTCOMES:
Perioperative blood loss | Hospital stay, from admission to third postoperative day.
  Measurement of loss (in mL), calculated with mathematical formulas proposed by Nadler and Good

SECONDARY OUTCOMES:
Blood transfusion rate | Hospital stay, from admission to third postoperative day
  Number of patients needing blood transfusion
Infection rate | 90 postoperative days
  Number of patients with surgical or medical infections (wound, pneumonia, urinary tract)
Thrombotic event rate | 90 postoperative days.
  Number of patients with postoperative thrombotic event (Deep Venous Thrombosis, Pulmonary Embolism, Myocardial Infarction, Stroke)

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Lizaur Utrilla, MD, Principal Investigator — Orthopaedic Surgery Department, Elda University Hospital
Locations (1):
- Elda University Hospital, Elda, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No